CLINICAL TRIAL: NCT05423899
Title: Humanoid Robot Intervention vs Treatment as Usual For Loneliness in Long-term Care Homes
Brief Title: Humanoid Robot vs Treatment as Usual for Loneliness
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn to due issues with insurance of the robot.
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Soham Rej MD, MSc, Principal Investigator, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 427283
Record Dates: First submitted 2022-06-01; First posted 2022-06-21 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-10

CONDITIONS: Loneliness; Depression; Stress; Anxiety; Quality of Life
Keywords: Loneliness; Humanoid Robot; Depression; Long-term Care; Stress
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Humanoid Robot (Experimental)
  Interventions: Behavioral: Grace Robot
- Treatment as Usual (Active Comparator)
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Grace Robot — The Grace robot was designed by Awakening Health/Hanson Robotics for healthcare settings and to interact with the elderly and those isolated by the COVID-19 pandemic. Grace is a robot with a human-like appearance, which can move, actively listen, engage in conversation and react appropriately to human emotions. Intervention activities will mostly consist of active listening and general discussions about topics of interest (e.g. hobbies, music). The participant will also have the option of other types of interactions with the robot, including robot-led meditation, robot-led light exercise, listening to music and singing. Because loneliness is a subjective experience and does not have a standardized solution, this is a personalized intervention approach. We anticipate that each older adult participant will have different needs and wishes when interacting with the robot, which will allow for a more natural interaction with the robot.
  Arms: Humanoid Robot
Behavioral: Treatment as Usual — The treatment as usual active control group will not receive the robot intervention. The investIgators have deliberately chosen the participating long-term care (LTC) homes due to their high frequency of social interactions for their clients as part of their routine care (e.g. one-on-one and group activities, family interaction, exercise groups) compared to most LTC homes settings, making TAU an active control.
  Arms: Treatment as Usual

SUMMARY:
The investigators are aiming to compare the effects of a humanoid robot intervention to treatment as usual, on loneliness and mental health outcomes in older adults living in long-term care, through an assessor-blinded randomized controlled trial.

DETAILED DESCRIPTION:
Seventy-four (n=74) older adults experiencing loneliness in 3 long-term care homes will be randomized 1:1 to an 8-week, twice a week social intervention with the Grace humanoid robot vs. a treatment as usual active control. The investigators will assess change (baseline to week 8) in (1) loneliness (primary outcome), (2) depression severity and (3) stress (secondary outcomes), as well as (4) other exploratory outcomes : anxiety, quality of life and reduction in acute healthcare utilization. The investigators will also assess the feasibility and acceptability of the intervention using qualitative methods.

ELIGIBILITY:
Inclusion Criteria:

* living in a LTC home setting in Montreal
* cognitively healthy, mild cognitive impairment (MCI) or mild dementia (MMSE score of >20/clinical opinion of LTC homes staff members)
* able to provide consent
* loneliness UCLA-3 score of ≥ 6 or more (moderate-severe loneliness).

Exclusion Criteria:

* do not speak English
* inability to provide consent
* moderate to severe dementia (MMSE score <18/diagnosis of moderate-severe dementia/clinical opinion of LTC homes staff members)
* significant hearing loss
* acutely unstable medical illnesses, including delirium, acute cerebrovascular/cardiovascular events within the last 6 months; having a terminal medical diagnosis with prognosis of less than 12 months
* high suicide risk (e.g. active suicidal ideation and/or current/recent intent or plan).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Change in the University of California Los Angeles 3-item Loneliness Scale | Baseline and Week 8
  Commonly-used validated scale to screen for loneliness. Higher scores on this scale mean higher levels of loneliness.

SECONDARY OUTCOMES:
Change in the Perceived Stress Scale | Baseline and Week 8
  14-item scale used to measure the degree to which life events are experienced and appraised as stressful. Higher scores on this scale mean higher stress levels.
Patient Health Questionnaire | Baseline and Week 8
  9-item self-report questionnaire used to diagnose depression and assess symptom severity. Higher scores on this scale mean more symptoms of depression.

OTHER OUTCOMES:
Generalized Anxiety Disorder-7 | Baseline and Week 8
  Commonly-used validated scale to measure anxiety. Higher scores on this scale mean more symptoms of anxiety.
EuroQoL-5 Dimensions | Baseline and Week 8
  Commonly-used validated scale to measure quality of life. Higher scores on this scale mean a better quality of life.
Change in acute healthcare utilization | Baseline and Week 8
  Number of hospitalizations and emergency room visits between baseline and primary intervention endpoint.

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plan

REFERENCES:
- [Derived] Lavin P, Lesage M, Monroe E, Kanevsky M, Gruber J, Cinalioglu K, Rej S, Sekhon H. Humanoid robot intervention vs. treatment as usual for loneliness in long-term care homes: Study protocol for a pilot randomized controlled trial. Front Psychiatry. 2022 Oct 21;13:1003881. doi: 10.3389/fpsyt.2022.1003881. eCollection 2022. PMID 36339874